CLINICAL TRIAL: NCT06796049
Title: Role of Behavioral Nudge as a Tool to Increase CRC Screening at an Urban Center Outpatient Clinic
Brief Title: Behavioral Nudge in Colorectal Cancer Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-00165
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Improving Fecal Immunochemical Test (FIT) Completion Rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time Period 1 (No Intervention): A FIT test is ordered by the provider and a patient care assistant (PCA) gives patient a FIT kit, which includes a specimen cup and instructions on how to use it, at the end of the visit prior to their departure.
- Time Period 2 (Experimental): A new information pamphlet is given to participants alongside the FIT kit at the end of the visit. The pamphlet contains an easy-to-read description of FIT screening adapted from the NYC department of health C5 Colorectal cancer (CRC) screening coalition pamphlet and lead-time CRC screening messaging tool, instructions on how to complete the test and the importance of FIT screening.
  Interventions: Behavioral: Information pamphlet
- Time Period 3 (Experimental): A new information pamphlet is given to participants along the FIT kit similar to "Time period 2", but includes a social norm driver in the pamphlet that displays the sub-par screening rate of our clinic compared to a collective New York State screening rate and a national screening rate goal set by the Centers for Disease Control and Prevention (CDC).
  Interventions: Behavioral: Information pamphlet + social norm driver

INTERVENTIONS:
Behavioral: Information pamphlet + social norm driver — The information pamphlet is given to participants at the end of the visit. The pamphlet contains an easy-to-read description of FIT screening adapted from the NYC department of health C5 Colorectal cancer (CRC) screening coalition pamphlet and lead-time CRC screening messaging tool, instructions on how to complete the test and the importance of FIT screening.
  The information pamphlet will also contain a social norm driver that displays the sub-par screening rate the clinic compared to a collective New York State screening rate and a national screening rate goal set by the CDC.
  Arms: Time Period 3
Behavioral: Information pamphlet — The information pamphlet is given to participants at the end of the visit. The pamphlet contains an easy-to-read description of FIT screening adapted from the NYC department of health C5 CRC screening coalition pamphlet and lead-time CRC screening messaging tool, instructions on how to complete the test and the importance of FIT screening.
  Arms: Time Period 2

SUMMARY:
The purpose of this study is to evaluate if a behavioral nudge principle known as social norm driver can be implemented to improve fecal immunochemical test (FIT) completion rates for patients' age 45-75 years old due for colorectal cancer screening at Bellevue Hospital Medicine Ambulatory Care Clinic. The study's endpoints include FIT screening completion rate and timeliness. Secondary analysis will look at demographic information such as age group, gender, prior screening, number of prior visits at the clinic.

ELIGIBILITY:
Time Period 1 Inclusion Criteria:

1. Patient at Bellevue Ambulatory Care Medicine Clinic between 1/1/2024 and 7/1/2024
2. Age 45-75 years old

Time Period 2 Inclusion Criteria:

1. Patient at Bellevue Ambulatory Care Resident Clinic
2. Age 45-75 years old
3. Has not had a FIT test within the past year
4. Can read either English or Spanish
5. Is able and willing to provide consent

Time Period 3 Inclusion Criteria:

1. Patient at Bellevue Ambulatory Care Resident Clinic
2. Age 45-75 years old
3. Has not had a FIT test completed within the past year
4. Can read either English or Spanish
5. Is able and willing to provide consent

Time Period 1 Exclusion Criteria:

1. Patient at a clinic that is not Bellevue Ambulatory Care Resident Clinic
2. Age outside of 45-75 years old

Time Period 2 Exclusion Criteria:

1. Patient at a clinic that is not Bellevue Ambulatory Care Resident Clinic
2. Age outside of 45-75 years old
3. Has had a FIT test completed within the past year
4. Cannot read either English or Spanish

Time Period 3 Exclusion Criteria:

1. Patient at a clinic that is not Bellevue Ambulatory Care Resident Clinic
2. Age outside of 45-75 years old
3. Has had a FIT test completed within the past year
4. Cannot read either English or Spanish

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time until the fecal immunochemical test (FIT) is returned to the clinic for processing | Month 3
  Study participants will be tracked for completion of their FIT screening test up until 3 months after the initial stool study was given.
Percentage of participants who completed the FIT screening test | Month 3
  Study participants will be tracked for completion of their FIT screening test up until 3 months after the initial stool study was given.

CONTACTS AND LOCATIONS:
Overall Officials: Aasma Shaukat, MD, Study Director — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be available to other researchers. Access to this aggregated study database will be limited to HIPAA certified investigators who have been IRB-approved for participation in this study.